CLINICAL TRIAL: NCT05309863
Title: Comparison Between the Efficacy of Residential and Ambulatory Weight Loss Programs for Pediatric Non-alcoholic Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-05660
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; Liver fibrosis; Lifestyle management; Multidisciplinary treatment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residential treatment: Patients administered for residential treatment of severe obesity will be included. Patients are treated according to standard of care in a multimodal program, focusing on increasing the level of physical activity, dietary intervention, acquiring healthy eating habits, and psychological support. Residential treatment is possible for a duration of maximum 1 year.
  Interventions: Behavioral: Lifestyle management
- Ambulatory treatment: Patients in specific pediatric obesity care pathways will be included. Patients are treated according to standard of care in a multimodal ambulatory program focusing on increasing the level of physical activity, dietary intervention, acquiring healthy eating habits, and psychological support.
  Interventions: Behavioral: Lifestyle management

INTERVENTIONS:
Behavioral: Lifestyle management — Increasing the level of physical activity, dietary intervention, acquiring healthy eating habits, and psychological support.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has become the most prevalent chronic liver disease worldwide, paralleling the obesity pandemic. Secondary to increasing rates of obesity in children and adolescents, the prevalence of NAFLD has more than doubled in the last decades and is now the most common pediatric liver disease.

At present, lifestyle modification by dietary intervention and increasing physical activity is the mainstay of treatment for pediatric NAFLD. Several studies have shown that lifestyle intervention and weight loss improve non-invasive markers of NAFLD. To the investigator's knowledge, data on fibrosis regression following lifestyle treatment in children and adolescents were lacking. The investigators therefore performed a prospective cohort study to investigate the impact of residential lifestyle treatment on liver steatosis and fibrosis in obese children and adolescents.

As a follow-up, the investigators now aim to compare these findings with a cohort of well-characterized patients undergoing multidisciplinary, yet ambulatory, weight loss treatment. As such, the investigators will compare the outcomes in two prospective patient cohorts in this non-randomized observational study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the lifestyle management program for obesity in one of the participating centres

Exclusion Criteria:

* Syndromic obesity
* Evidence of liver disease of other causes (viral, auto-immune, genetic)
* Average daily alcohol consumption of >20g/day
* Unvalid screening Fibroscan
* Treatment with drugs which can induce liver steatosis or fibrosis (e.g. systemic corticosteroids, methotrexate)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with obesity (BMI higher than the 95th weight percentile)
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver fibrosis | 6 months of lifestyle intervention
  Liver fibrosis will be quantified using Fibroscan, and patients will be divided into disease stages based on published cut-offs.

SECONDARY OUTCOMES:
Improvement of liver fibrosis | 12 months of lifestyle intervention
  Liver fibrosis will be quantified using Fibroscan, and patients will be divided into disease stages based on published cut-offs.
Improvement of liver steatosis | 6 months of lifestyle intervention
  Liver steatosis will be quantified using controlled attenuation parameter on the Fibroscan
Improvement of liver steatosis | 12 months of lifestyle intervention
  Liver steatosis will be quantified using controlled attenuation parameter on the Fibroscan
Resolution of liver steatosis | 6 months of lifestyle intervention
  Liver steatosis will be quantified using controlled attenuation parameter on the Fibroscan. Resolution of steatosis is identified as CAP <248 dB/m at follow-up in patients with baseline CAP of 248 dB/m or higher.
Resolution of liver steatosis | 12 months of lifestyle intervention
  Liver steatosis will be quantified using controlled attenuation parameter on the Fibroscan. Resolution of steatosis is identified as CAP <248 dB/m at follow-up in patients with baseline CAP of 248 dB/m or higher.
Resolution of liver fibrosis | 6 months of lifestyle intervention
  Liver fibrosis will be quantified using Fibroscan. Resolution of fibrosis is identified as liver stiffness <7.0 kPa at follow-up in patients with baseline liver stiffness of 7.0 kPa or higher.
Resolution of liver fibrosis | 12 months of lifestyle intervention
  Liver fibrosis will be quantified using Fibroscan. Resolution of fibrosis is identified as liver stiffness <7.0 kPa at follow-up in patients with baseline liver stiffness of 7.0 kPa or higher.
Improvement in ALT | 6 months of lifestyle intervention
  Proportion of patients with at least 30% decrease in serum ALT levels at follow-up, out of the patients with baseline elevated ALT
Improvement in ALT | 12 months of lifestyle intervention
  Proportion of patients with at least 30% decrease in serum ALT levels at follow-up, out of the patients with baseline elevated ALT

CONTACTS AND LOCATIONS:
Overall Officials: Ruth De Bruyne, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - AZ Jan Palfijn, Ghent, East-Flanders
  - University Hospital Gent, Ghent, East-Flanders
  - Zeepreventorium, De Haan, West-Flanders

IPD SHARING:
Plan to Share IPD: Undecided
The plan can be obtained by contacting the researchers with a worked-out protocol for study in which these data can be used.

REFERENCES:
- [Background] Lefere S, Dupont E, De Guchtenaere A, Van Biervliet S, Vande Velde S, Verhelst X, Devisscher L, Van Vlierberghe H, Geerts A, De Bruyne R. Intensive Lifestyle Management Improves Steatosis and Fibrosis in Pediatric Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2022 Oct;20(10):2317-2326.e4. doi: 10.1016/j.cgh.2021.11.039. Epub 2021 Dec 4. PMID 34871812
- [Background] Nobili V, Vizzutti F, Arena U, Abraldes JG, Marra F, Pietrobattista A, Fruhwirth R, Marcellini M, Pinzani M. Accuracy and reproducibility of transient elastography for the diagnosis of fibrosis in pediatric nonalcoholic steatohepatitis. Hepatology. 2008 Aug;48(2):442-8. doi: 10.1002/hep.22376. PMID 18563842
- [Background] Ciardullo S, Monti T, Perseghin G. Prevalence of Liver Steatosis and Fibrosis Detected by Transient Elastography in Adolescents in the 2017-2018 National Health and Nutrition Examination Survey. Clin Gastroenterol Hepatol. 2021 Feb;19(2):384-390.e1. doi: 10.1016/j.cgh.2020.06.048. Epub 2020 Jul 3. PMID 32623006